CLINICAL TRIAL: NCT03523585
Title: A Phase 3, Multicenter, Randomized, Open-label, Active-controlled Study of Trastuzumab Deruxtecan (DS-8201a), an Anti-HER2-antibody Drug Conjugate, Versus Treatment of Investigator's Choice for HER2-positive, Unresectable and/or Metastatic Breast Cancer Subjects Previously Treated With T-DM1
Brief Title: DS-8201a in Pre-treated HER2 Breast Cancer That Cannot be Surgically Removed or Has Spread [DESTINY-Breast02]
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-U301; 2018-000221-31 (EudraCT Number); 184017 (Registry Identifier: JAPIC CTI); DESTINY-Breast02 (Other: Daiichi Sankyo and AstraZeneca)
Record Dates: First submitted 2018-04-13; First posted 2018-05-14 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic breast cancer; DS 8201a; DESTINY - Breast 02
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan; Capecitabine; Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Trastuzumab deruxtecan (DS-8201a) (Experimental): HER2 positive, unresectable and/or metastatic breast cancer participants previously treated with standard of care HER2 therapies, including ado-trastuzumab emtansine (T-DM1), randomized to treatment with DS-8201a
  Interventions: Drug: Trastuzumab deruxtecan
- Trastuzumab+capecitabine (Active Comparator): HER2 positive, unresectable and/or metastatic breast cancer participants previously treated with standard of care HER2 therapies, including ado-trastuzumab emtansine (T-DM1), randomized to investigator's choice treatment with Trastuzumab/capecitabine
  Interventions: Drug: Capecitabine; Drug: Trastuzumab
- Lapatinib+capecitabine (Active Comparator): HER2 positive, unresectable and/or metastatic breast cancer participants previously treated with standard of care HER2 therapies, including ado-trastuzumab emtansine (T-DM1), randomized to investigator's choice treatment with Lapatinib/capecitabine
  Interventions: Drug: Capecitabine; Drug: Lapatinib

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — DS-8201a is sterile lyophilized powder reconstituted into a sterile aqueous solution (100 mg/5 mL) to be administered as intravenous (IV) dose
  Other Names: DS-8201a; T-DXd
  Arms: Trastuzumab deruxtecan (DS-8201a)
Drug: Capecitabine — Investigator's choice Standard of Care when combined with trastuzumab or lapatinib
  Other Names: Investigator's Choice Comparative Therapy
  Arms: Lapatinib+capecitabine; Trastuzumab+capecitabine
Drug: Lapatinib — Investigator's choice Standard of Care when combined with capecitabine
  Other Names: Investigator's Choice Comparative Therapy
  Arms: Lapatinib+capecitabine
Drug: Trastuzumab — Investigator's choice Standard of Care when combined with capecitabine
  Other Names: Investigator's Choice Comparative Therapy
  Arms: Trastuzumab+capecitabine

SUMMARY:
This study will compare DS 8201a to standard treatment.

Participants must have HER2 breast cancer that has been treated before.

Their cancer:

* cannot be removed by an operation
* has spread to other parts of the body

DETAILED DESCRIPTION:
The study is designed to compare DS 8201a versus standard of care (investigator's choice) in subjects with unresectable and/or metastatic breast cancer previously treated with T-DM1.

ELIGIBILITY:
Inclusion Criteria:

* Is the age of majority in their country
* Has pathologically documented breast cancer that:

  1. is unresectable or metastatic
  2. has confirmed HER2-positive expression as determined according to American Society of Clinical Oncology - College of American Pathologists guidelines evaluated at a central laboratory
  3. was previously treated with ado-trastuzumab emtansine (T-DM1)
* Has documented radiologic progression (during or after most recent treatment or within 6 months after completing adjuvant therapy)
* Is HER2 positive as confirmed by central laboratory assessment of most recent tumor tissue sample available. If archived tissue is not available, agrees to provide a fresh biopsy.
* Male and female participants of reproductive/childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least:

  1. 7 months after the last dose of DS-8201a (females); 4.5 months after last dose of DS-8201a (males)
  2. 6 months after the last dose of lapatinib/capecitabine for female participants (3 months for male participants)
  3. 7 months after the last dose of trastuzumab/capecitabine
* Has adequate hematopoietic, renal and hepatic functions

Exclusion Criteria:

* Has previously participated in an antibody drug conjugate study sponsored by Daiichi Sankyo. Prior treatment in the adjuvant/neo-adjuvant setting would be allowed if progression of disease did not occur within 12 months of end of adjuvant therapy
* Has had prior treatment with capecitabine
* Has uncontrolled or significant cardiovascular disease
* Has a history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening
* Has active central nervous system (CNS) metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2026-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Global Team Leader, Study Director — Daiichi Sankyo
Locations (227):
- United States (41):
  - Ironwood Cancer Research Centers, Chandler, Arizona
  - UCLA Hematology Oncology - Main Site, Los Angeles, California
  - Pacific Cancer Care, Monterey, California
  - Sharp Memorial Hospital, San Diego, California
  - Innovative Clinical Research Institute, Whittier, California
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Florida Cancer Specialists-Broadway, Fort Myers, Florida
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children/Univ of HI, Honolulu, Hawaii
  - Loyola University Health System, Maywood, Illinois
  - Community Hospital, Munster, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Cornell-Beshore Cancer Institute, Joplin, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Health Midwest Ventures Group, Inc d/b/a HCA MidAmerica Division, LLC, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - North Shore Hematology Oncology Associates, PC, East Setauket, New York
  - Memorial Sloan-Kettering Cancer Center (MSKCC) - New York, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Dayton Physicians, LLC, Kettering, Ohio
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC Chattanooga, Chattanooga, Tennessee
  - The West Clinic, Germantown, Tennessee
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
- Australia (16):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Macquarie University Hospital, Sydney, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Peninsula and South Eastern Haematology & Oncology Group, Frankston, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sunshine Hospital, Saint Albans, Victoria
  - South West Oncology, Warrnambool, Victoria
  - Ballarat Oncology & Haematology Service, Wendouree, Victoria
  - St John of God Subiaco Hospital, Subiaco, Western Australia
  - Calvary North Adelaide Hospital, Bruce
- Belgium (6):
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Maria Middelares, Ghent
  - Az Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU UCL Namur site de Sainte Elisabeth, Namur
- Brazil (14):
  - Pronutrir, Fortaleza, Ceará
  - NOB - Núcleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - AMO - Assistência Multidisciplinar em Oncologia, Salvador, Estado de Bahia
  - Oncobio Servicos de Saude, Nova Lima, Minas Gerais
  - HGB - Hospital Giovanni Battista - Mãe de Deus Center, Porto Alegre, Rio Grande do Sul
  - CliniOnco - Tratamento Integrado do Câncer, Porto Alegre, Rio Grande do Sul
  - Escosteguy Barrios, Carlos Henrique, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - Clínica de Neoplasias Litoral Ltda., Itajaí, Santa Catarina
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - IBCC - Instituto Brasileiro de Controle do Câncer, São Paulo, São Paulo
  - COI - Clínicas Oncológicas Integradas, Rio de Janeiro
  - Sociedade Beneficiente de Senhoras Hospital Sírio Libanês, São Paulo
  - A. C. Camargo Cancer Center, São Paulo
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice v Motole, Prague
  - Nemocnice Na Bulovce, Prague
- France (23):
  - Hôpital Nord - CHU Marseille, Marseille, Bouches-du-Rhône
  - Centre François Baclesse, Caen, Calvados
  - CARIO - Centre Armoricain de Radiothérapie, Imagerie médicale et Oncologie, Plérin, Cotes d'Armor
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - CHU Brest - Hôpital Morvan, Brest, Finistere
  - Hôpital Privé d'Antony, Antony, Hauts De Seine
  - Centre René Huguenin, Saint-Cloud, Hauts De Seine
  - Clinique Clementville, Montpellier, Herault
  - Institut Régional du Cancer de Montpellier, Montpellier, Herault
  - CRLCC Eugene Marquis, Rennes, Ille Et Vilaine
  - Centre Oscar Lambret, Lille, Nord
  - Centre de cancerologie les Dentellieres, Valenciennes, Nord
  - Institut Curie - site de Paris, Paris, Paris
  - Centre Hospitalier de la côte Basque, Bayonne, Pyrenees Atlantiques
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans, Sarthe
  - Centre Henri Becquerel, Rouen, Seine Maritime
  - Institut Sainte Catherine, Avignon, Vaculuse
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Institut Curie - site de Paris, Paris
  - Hopital Tenon, Paris
- Germany (11):
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Marienhospital Bottrop gGmbH, Bottrop, Rhineland-Palatinate
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck, Schleswig-Holstein
  - Helios-Kliniken Berlin-Buch, Berlin
  - Kliniken Koeln, Cologne
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Leipzig AoeR, Leipzig
  - Klinikum der Universitaet Muenchen - Campus Grosshardern, Munich
  - Universitaetsklinikum Muenster, Müenster
  - Haematologisch-Onkologische Schwerpunktpraxis, Troisdorf
- Greece (5):
  - 251 General Air Force Hospital, Athens
  - General Hospital of Athens "Alexandra", Athens
  - General Oncology Hospital of Kifissia " Agioi Anargyroi", Athens
  - University General Hospital of Heraklion, Heraklion
  - Euromedica General Clinic Thessaloniki, Thessaloniki
- Israel (7):
  - Rambam Health Care Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Sapir Medical Center, Meir Hospital, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (19):
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), Monza, Milano
  - IRCCS Centro di Riferimento Oncologico, Aviano, Pordenone
  - Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Cona
  - Istituto Nazionale per la Ricerca sul Cancro di Genova, Genova
  - Azienda Ospealiera della Provincia di Lecco, Lecco
  - Azienda Ospedaliera Ospedali Riuniti Papardo-Piemonte, Messina
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - A.O.U. Policlinico di Modena, Modena
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Japan (23):
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Kindai University Hospital, Ōsakasayama-shi, Osaka
  - National Cancer Center Hospital, Chūōku, Tokyo-To
  - NHO Shikoku Cancer Center, Ehime
  - NHO Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - NHO Hokkaido Cancer Center, Hokkaido
  - Hyōgo College of Medicine Hospital, Hyōgo
  - St. Marianna University School of Medicine Hospital, Kanagawa
  - Kanagawa Cancer Center, Kanagawa
  - Kyoto University Hospital, Kyoto
  - Tohoku University Hospital, Miyagi
  - Aichi Cancer Center Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - NHO Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - Toranomon Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Tokyo Medical University Hospital, Tokyo
- South Korea (13):
  - Inha University Hospital, Incheon, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (20):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Especialidades de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Infanta Cristina, Badajoz
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano de Oncologia IVO, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Turkey (Türkiye) (16):
  - Acibadem Adana Hospital, Adana
  - Adana Numune Training and Research Hospital, Adana
  - Ankara Yildirim Beyazit Uni. Med. Fac.Ankara City Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Uludag University Medical Faculty, Bursa
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Bakirkoy Dr. Sadi Konuk Teaching and Research Hospital, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - Medical Park Goztepe Hospital, Istanbul
  - Istanbul Medeniyet Uni Goztepe Training & Research Hospital, Istanbul
  - Kartal Lutfi Kirdar Research and Training Hospital, Istanbul
  - Izmir Medicalpark Hospital, Izmir
  - Konya Necmettin Erbakan University Meram Faculty of Medicine, Konya
  - Sakarya Traning and Research Hospital, Sakarya
  - Medical Park Samsun Hastanesi, Samsun
  - Namik Kemal University, Tekirdağ
- United Kingdom (9):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - Derriford Hospital, Plymouth, Devon
  - Aberdeen Royal Infirmary, Aberdeen, Grampian Region
  - Queen Mary University of London, London, Greater London
  - University College London Hospitals, London, Greater London
  - Sarah Cannon Research Institute UK, London, Greater London
  - Western General Hospital, Edinburgh, Lothian Region
  - Nottingham University Hospitals City Campus, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Result] Andre F, Hee Park Y, Kim SB, Takano T, Im SA, Borges G, Lima JP, Aksoy S, Gavila Gregori J, De Laurentiis M, Bianchini G, Roylance R, Miyoshi Y, Armstrong A, Sinha R, Ruiz Borrego M, Lim E, Ettl J, Yerushalmi R, Zagouri F, Duhoux FP, Fehm T, Gambhire D, Cathcart J, Wu C, Chu C, Egorov A, Krop I. Trastuzumab deruxtecan versus treatment of physician's choice in patients with HER2-positive metastatic breast cancer (DESTINY-Breast02): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2023 May 27;401(10390):1773-1785. doi: 10.1016/S0140-6736(23)00725-0. Epub 2023 Apr 20. PMID 37086745
- [Result] Fehm T, Cottone F, Dunton K, Andre F, Krop I, Park YH, De Laurentiis M, Miyoshi Y, Armstrong A, Borrego MR, Yerushalmi R, Duhoux FP, Takano T, Lu W, Egorov A, Kim SB. Trastuzumab deruxtecan versus treatment of physician's choice in patients with HER2-positive metastatic breast cancer (DESTINY-Breast02): patient-reported outcomes from a randomised, open-label, multicentre, phase 3 trial. Lancet Oncol. 2024 May;25(5):614-625. doi: 10.1016/S1470-2045(24)00128-1. PMID 38697155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 608 participants were enrolled at study sites in 15 countries. Primary results reported is from first participant randomized up to data cut-off date of 30 Jun 2022. The results presented are based on primary analysis up to 46 months.
Pre-assignment Details: Participants in The Physician's Choice (TPC) group were randomized to 1 of the following 2 regimens: trastuzumab/capecitabine or lapatinib/capecitabine. As prespecified in the protocol, participants were assessed and reported separately per comparator arm for the disposition, baseline characteristics, and safety tables. For efficacy assessments, all participants in the TPC group were combined and assessed together.
Groups:
- Trastuzumab Deruxtecan (T-DXd): Participants with HER2 positive, unresectable and/or metastatic breast cancer participants previously treated with standard of care HER2 therapies, including ado-trastuzumab emtansine (T-DM1), who received T-DXd as a sterile intravenous (IV) solution at a dose of 5.4 mg/kg every 3 weeks (Q3W).
- Trastuzumab+Capecitabine: Participants with HER2 positive, unresectable and/or metastatic breast cancer participants previously treated with standard of care HER2 therapies, including ado-trastuzumab emtansine (T-DM1), who received investigator's choice treatment, Trastuzumab/Capecitabine.
- Lapatinib+Capecitabine: Participants with HER2 positive, unresectable and/or metastatic breast cancer participants previously treated with standard of care HER2 therapies, including ado-trastuzumab emtansine (T-DM1), who received investigator's choice treatment, Lapatinib/Capecitabine.
Period: Overall Study
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Trastuzumab+Capecitabine | Lapatinib+Capecitabine
Started | 406 | 91 | 111
Randomized | 406 | 91 | 111
Randomized But Not Treated | 2 | 4 | 3
Completed (Completed = Participants who are on-going study treatment as of 30 Jun 22, Not Completed = Participants who discontinued treatment and participants randomized but not treated.) | 94 | 1 | 4
Not Completed | 312 | 90 | 107
Not completed — Progressive Disease | 174 | 64 | 77
Not completed — Adverse Event | 74 | 5 | 9
Not completed — Withdrawal by Subject | 30 | 11 | 6
Not completed — Clinical Progression | 23 | 5 | 10
Not completed — Death | 4 | 0 | 1
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Miscellaneous | 1 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 1
Not completed — Randomized But Not Treated | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Trastuzumab+Capecitabine | Lapatinib+Capecitabine | Total
Number analyzed (Participants) | 406 | 91 | 111 | 608
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 321 | 73 | 91 | 485
  >=65 years | 85 | 18 | 20 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (11.99) | 55.7 (11.40) | 54.6 (11.06) | 54.8 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 403 | 89 | 111 | 603
  Male | 3 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 122 | 20 | 36 | 178
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 10 | 2 | 5 | 17
  White | 257 | 66 | 61 | 384
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 15 | 3 | 8 | 26
Region of Enrollment [Number; unit: participants]
  United States | 41 | 14 | 9 | 64
  Czechia | 1 | 2 | 0 | 3
  Japan | 46 | 6 | 18 | 70
  United Kingdom | 27 | 4 | 4 | 35
  Spain | 29 | 8 | 7 | 44
  Greece | 9 | 3 | 2 | 14
  South Korea | 66 | 11 | 17 | 94
  Turkey | 36 | 12 | 4 | 52
  Belgium | 4 | 1 | 0 | 5
  Brazil | 41 | 10 | 8 | 59
  Italy | 33 | 3 | 17 | 53
  Israel | 14 | 0 | 4 | 18
  France | 37 | 8 | 12 | 57
  Australia | 10 | 7 | 4 | 21
  Germany | 12 | 2 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Based on Blinded Independent Central Review (BICR) in Participants With HER2-positive, Unresectable and/or Metastatic Breast Cancer Participants Previously Treated With Trastuzumab Emtansine
Description: Progression-free survival (PFS) by BICR was defined as the time from the date of randomization to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause.
Time Frame: Baseline up to 46 months postdose
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set at data cut-off date of 30 Jun 2022.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment of Investigator's/Physician's Choice (TPC): Participants with HER2 positive, unresectable and/or metastatic breast cancer participants previously treated with standard of care HER2 therapies, including ado-trastuzumab emtansine (T-DM1), who received investigator's choice treatment, Trastuzumab/Capecitabine or Lapatinib/Capecitabine.
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Treatment of Investigator's/Physician's Choice (TPC)
Number analyzed (Participants) | 406 | 202
months | 17.8 [14.3 to 20.8] | 6.9 [5.5 to 8.4]
Statistical Analysis 1: Comparison: Trastuzumab Deruxtecan (T-DXd) vs Treatment of Investigator's/Physician's Choice (TPC); Test type: Superiority; p < 0.000001, Log Rank — Stratified Log-rank p-value; p value based on log-rank stratified by hormone receptor status, prior treatment with pertuzumab, and history of visceral disease, as defined by IXRS; Hazard Ratio (HR) = 0.3589, 95% CI 2-sided [0.2840 to 0.4535] — Hazard Ratio based on stratified Cox proportional hazards model with stratification factors: hormone receptor status, prior treatment with pertuzumab, and history of visceral disease, as defined by the IXRS

2. Secondary Outcome: Overall Survival (OS) in Participants With HER2-positive, Unresectable and/or Metastatic Breast Cancer Participants Previously Treated With Trastuzumab Emtansine
Description: Overall survival (OS) was defined as the time from the date of randomization to the date of death due to any cause. If there is no death reported for a subject before the data cutoff for OS analysis, OS will be censored at the last contact date at which the subject is known to be alive.
Time Frame: Baseline up to 46 months postdose
Population: Overall survival (OS) was assessed in the Full Analysis Set at data cut-off date of 30 Jun 2022.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Treatment of Investigator's/Physician's Choice (TPC)
Number analyzed (Participants) | 406 | 202
months | 39.2 [32.7 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. | 26.5 [21.0 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to insufficient number of events.
Statistical Analysis 1: Comparison: Trastuzumab Deruxtecan (T-DXd) vs Treatment of Investigator's/Physician's Choice (TPC); Test type: Superiority; p = 0.0021, Log Rank — Stratified Log-rank p-value; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.6575, 95% CI 2-sided [0.5023 to 0.8605] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR) in Participants With HER2-positive, Unresectable and/or Metastatic Breast Cancer Participants Previously Treated With Trastuzumab Emtansine
Description: The Objective Response Rate (ORR) was defined as the percentage of participants who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), assessed by BICR and investigator assessment based on RECIST version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Confirmed ORR based on BICR and Investigator Assessment is reported.
Time Frame: Baseline up to 46 months postdose
Population: Objective response rate (ORR) was assessed in the Full Analysis Set at data cut-off date of 30 Jun 2022.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Treatment of Investigator's/Physician's Choice (TPC)
Number analyzed (Participants) | 406 | 202
Percentage of Participants
  BICR | 69.7 [65.0 to 74.1] | 29.2 [23.0 to 36.0]
  Investigator Assessment | 74.1 [69.6 to 78.3] | 26.7 [20.8 to 33.4]
Statistical Analysis 1: Comparison: Trastuzumab Deruxtecan (T-DXd) vs Treatment of Investigator's/Physician's Choice (TPC); Statistical Analysis for BICR Assessment; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test adjusted for stratification factors: hormone receptor status, prior treatment with pertuzumab, and history of visceral disease, as defined by the IXRS
Statistical Analysis 2: Comparison: Trastuzumab Deruxtecan (T-DXd) vs Treatment of Investigator's/Physician's Choice (TPC); Statistical Analysis for Investigator Assessment; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Duration of Response (DoR) Based on BICR in Participants With HER2-positive, Unresectable and/or Metastatic Breast Cancer Participants Previously Treated With Trastuzumab Emtansine
Description: Duration of Response (DoR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause. DoR in participants with confirmed CR/PR based on BICR and investigator assessment is reported.
Time Frame: Baseline up to 46 months postdose
Population: Duration of Response (DoR) was assessed in the Full Analysis Set of participants with confirmed CR/PR at data cut-off date of 30 Jun 2022.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Treatment of Investigator's/Physician's Choice (TPC)
Number analyzed (Participants) | 283 | 59
months | 19.6 [15.9 to NA] — Upper CI was not estimable due to insufficient number of events. | 8.3 [5.8 to 9.5]

5. Secondary Outcome: Progression-Free Survival (PFS) Based on Investigator Assessment in Participants With HER2-positive, Unresectable and/or Metastatic Breast Cancer Participants Previously Treated With Trastuzumab Emtansine
Description: Progression-free survival (PFS) by investigator assessment was defined as the time from the date of randomization to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause.
Time Frame: Up to 46 months
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set at data cut-off date of 30 Jun 2022.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Treatment of Investigator's/Physician's Choice (TPC)
Number analyzed (Participants) | 406 | 202
months | 16.7 [14.3 to 19.6] | 5.5 [4.4 to 7.0]
Statistical Analysis 1: Comparison: Trastuzumab Deruxtecan (T-DXd) vs Treatment of Investigator's/Physician's Choice (TPC); Test type: Superiority; p < 0.000001, Log Rank — Stratified Log-rank p-value; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.2828, 95% CI 2-sided [0.2270 to 0.3524] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up to 47 days after last dose of the study drug, up 46 months.
Description: A Treatment-emergent adverse event (TEAE) is defined as an AE that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the initiating the study drug until 47 days after last dose of the study drug. Adverse Events were assessed in the Safety Analysis Set at data cut-off date of 30 Jun 2022. All-Cause Mortality was analyzed in the Full Analysis Set. Serious and Other Adverse Events were analyzed in the Safety Analysis Set.
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Trastuzumab+Capecitabine | Lapatinib+Capecitabine
All-Cause Mortality (participants affected / at risk) | 143/406 | 40/91 | 46/111
Serious Adverse Events (participants affected / at risk) | 103/404 | 19/87 | 27/108
Other Adverse Events (participants affected / at risk) | 398/404 | 79/87 | 102/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Deruxtecan (T-DXd) (N=404) | Trastuzumab+Capecitabine (N=87) | Lapatinib+Capecitabine (N=108)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Stress Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Autoimmune Thyroiditis (Cardiac disorders) | 1 | 0 | 0
Autoimmune Thyroiditis (Endocrine disorders) | 1 | 0 | 0
Scleritis (Eye disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 3 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 0
Asthenia (General disorders) | 2 | 0 | 0
Disease Progression (General disorders) | 1 | 1 | 3
General Physical Health Deterioration (General disorders) | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 1
Covid-19 (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 6 | 0 | 1
Covid-19 Pneumonia (Infections and infestations) | 2 | 0 | 0
Device Related Infection (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 2 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 1
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0
Post Procedural Infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 0
Radiation Necrosis (Injury, poisoning and procedural complications) | 2 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases To Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pulmonary Tumour Thrombotic Microangiopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain Oedema (Nervous system disorders) | 2 | 0 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0
Monoplegia (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Vasogenic Cerebral Oedema (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0
Breast Pain (Reproductive system and breast disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Brachiocephalic Vein Thrombosis (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Sepsis (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1
Gastric Antral Vascular Ectasia (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis Bacterial (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1
Pancreatic Enzymes Increased (Investigations) | 0 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertensive Urgency (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Deruxtecan (T-DXd) (N=404) | Trastuzumab+Capecitabine (N=87) | Lapatinib+Capecitabine (N=108)
Anaemia (Blood and lymphatic system disorders) | 114 | 13 | 13
Neutropenia (Blood and lymphatic system disorders) | 65 | 4 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 41 | 4 | 7
Leukopenia (Blood and lymphatic system disorders) | 23 | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 21 | 1 | 1
Dry Eye (Eye disorders) | 23 | 4 | 5
Nausea (Gastrointestinal disorders) | 292 | 29 | 44
Vomiting (Gastrointestinal disorders) | 150 | 9 | 14
Constipation (Gastrointestinal disorders) | 142 | 12 | 9
Diarrhoea (Gastrointestinal disorders) | 109 | 33 | 69
Dyspepsia (Gastrointestinal disorders) | 48 | 6 | 12
Abdominal Pain (Gastrointestinal disorders) | 45 | 7 | 11
Stomatitis (Gastrointestinal disorders) | 44 | 11 | 25
Abdominal Pain Upper (Gastrointestinal disorders) | 38 | 7 | 11
Fatigue (General disorders) | 144 | 20 | 32
Asthenia (General disorders) | 97 | 6 | 13
Pyrexia (General disorders) | 51 | 5 | 7
Oedema Peripheral (General disorders) | 27 | 4 | 5
Mucosal Inflammation (General disorders) | 15 | 6 | 9
Covid-19 (Infections and infestations) | 47 | 1 | 2
Urinary Tract Infection (Infections and infestations) | 34 | 3 | 3
Nasopharyngitis (Infections and infestations) | 21 | 3 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 21 | 3 | 3
Paronychia (Infections and infestations) | 10 | 3 | 11
Neutrophil Count Decreased (Investigations) | 79 | 7 | 7
Weight Decreased (Investigations) | 71 | 2 | 5
Aspartate Aminotransferase Increased (Investigations) | 66 | 5 | 18
Alanine Aminotransferase Increased (Investigations) | 61 | 6 | 14
White Blood Cell Count Decreased (Investigations) | 59 | 5 | 4
Platelet Count Decreased (Investigations) | 49 | 5 | 7
Lymphocyte Count Decreased (Investigations) | 30 | 2 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 24 | 4 | 4
Blood Bilirubin Increased (Investigations) | 20 | 4 | 17
Decreased Appetite (Metabolism and nutrition disorders) | 124 | 15 | 20
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 | 7 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 36 | 1 | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 24 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 4 | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 13 | 4 | 7
Headache (Nervous system disorders) | 79 | 7 | 5
Dysgeusia (Nervous system disorders) | 33 | 3 | 1
Dizziness (Nervous system disorders) | 32 | 5 | 9
Neuropathy Peripheral (Nervous system disorders) | 12 | 6 | 4
Insomnia (Psychiatric disorders) | 25 | 6 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 53 | 7 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 3 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 33 | 5 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 25 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 150 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 27 | 3 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 2 | 6
Dry Skin (Skin and subcutaneous tissue disorders) | 11 | 3 | 6
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 7 | 48 | 52
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 6 | 2 | 6
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 10
Skin Toxicity (Skin and subcutaneous tissue disorders) | 1 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT03523585/Prot_SAP_001.pdf